CLINICAL TRIAL: NCT01511783
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of E2609 in Healthy Subjects
Brief Title: Evaluation of the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of E2609 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2609-A001-002
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- E2609 (Experimental): E2609 at ascending doses
  Interventions: Drug: E2609
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2609 — E2609 to be administered for 14 days, concurrently with placebo controls. Doses will be 25, 50, and 200 mg once daily by the oral route, each dose administered to a separate cohort (group) of subjects. After each dose has been administered to all subjects in a given cohort, safety and tolerability findings will be evaluated and a decision made by the sponsor and investigators as to whether or not to proceed to the next higher dose.
  Arms: E2609
Drug: Placebo — E2609 to be administered for 14 days, concurrently with placebo controls. Doses will be 25, 50, and 200 mg once daily by the oral route, each dose administered to a separate cohort (group) of subjects. After each dose has been administered to all subjects in a given cohort, safety and tolerability findings will be evaluated and a decision made by the sponsor and investigators as to whether or not to proceed to the next higher dose.
  Arms: Placebo

SUMMARY:
The purpose of this single-center, randomized, double-blind, placebo-controlled, study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of E2609 when administered to healthy elderly subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males and females
* Female subjects must be of non-childbearing potential
* Aged 50 to 85 years, inclusive BMI of 18 to 32 kg/m2 at screening
* Thyroid function tests within normal rangeMini-Mental State Examination score of 28-30, inclusive

Key Exclusion Criteria:

* History of neurological abnormalities, including seizures
* Any clinically significant abnormality of the ECG at Screening and Baseline including QTc prolongation
* History of ischemic heart disease, cardiac arrhythmias, cerebrovascular diseases
* Other medical conditions that are not stably controlled
* Presence of orthostatic hypotension

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 19 days

SECONDARY OUTCOMES:
Plasma Cmax and AUC (0-24h) of E2609 on Day 1 and Day 14 | 20 days
Plasma Aβ(1-x) Amax (defined as maximum change (%) of E2609 levels compared to time-matched baseline at a single time point within 24 hours postdose) in plasma and cerebrospinal fluid, plasma and CSF | 20 days
Time at which Amax occurs for plasma Aβ(1-x) | 20 days
Area under the plasma Aβ(1-x) concentration, AUAC(0-24h), by time curve from time 0 to time 24 hours on Day -1, Day 1, and Day 14 | 20 days
Change (%) in plasma Aβ(1-x) AUAC within 24 hours comparing Day 1 to Day -1 and Day 14 to Day -1 | 20 days
Percent change of Aβ(1-x) in CSF from Day -2 to Day 14 | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Craig Curtis, Principal Investigator — Compass Research Phase 1, LLC
Locations (1):
- Compass Research Phase 1, LLC, Orlando, Florida, United States